CLINICAL TRIAL: NCT06522555
Title: The Efficacy and Safety of Pola-ZR2 (Polatuzumab Vedotin, Zanubrutinib, Rituximab and Lenalidomide) Versus ZR2 (Zanubrutinib, Rituximab and Lenalidomide) in the Treatment of Old Patients With de Novo Diffuse Large B-cell Lymphoma: A Multicenter, Prospective, Randomized, Open-label, Controlled Trial
Brief Title: The Efficacy and Safety of Pola-ZR2 Versus ZR2 in the Treatment of Old Patients With de Novo Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director, Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POTENT STUDY
Record Dates: First submitted 2024-07-07; First posted 2024-07-26 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: diffuse large B-cell lymphoma; polatuzumab vedotin; zanubrutinib; lenalidomide; rituximab; old patients; unfit; frail
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; zanubrutinib; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pola-ZR2 (Experimental): six courses of polatuzumab vedotin, zanubrutinib, rituximab and lenalidomide induction therapy and lenalidomide maintenance therapy
  Interventions: Drug: polatuzumab vedotin, zanubrutinib, rituximab and lenalidomide
- ZR2 (Active Comparator): six courses of zanubrutinib, rituximab and lenalidomide induction therapy and lenalidomide maintenance therapy
  Interventions: Drug: zanubrutinib, rituximab and lenalidomide

INTERVENTIONS:
Drug: polatuzumab vedotin, zanubrutinib, rituximab and lenalidomide — Drug: Polatuzumab vedotin, Zanubrutinib, Lenalidomide and Rituximab (Pola-ZR2)
  Induction therapy:
  The Pola-ZR2 regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 21 days. Participants will receive a total of 6 cycles.
  Dosage:
  Polatuzumab vedotin 1.8 mg/kg, day 2 on the 1st cycle and day 1 on the 2nd to 6th cycle; Zanubrutinib, 160 mg bid, po, day 1-21; Lenalidomide, 25 mg qd, po, day 2-11; Rituximab, 375 mg/m2, ivgtt, day 1.
  Maintenance therapy:
  Patients who receive complete response or partial response after induction therapy will receive lenalidomide 25 mg qd po during 1-10 days in every 21 days for 2 years.
  Arms: Pola-ZR2
Drug: zanubrutinib, rituximab and lenalidomide — Drug: Zanubrutinib, Lenalidomide and Rituximab (ZR2)
  Induction therapy:
  The ZR2 regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 21 days. Participants will receive a total of 6 cycles.
  Dosage:
  Zanubrutinib, 160 mg bid, po, day 1-21; Lenalidomide, 25 mg qd, po, day 2-11; Rituximab, 375 mg/m2, ivgtt, day 1.
  Maintenance therapy:
  Patients who receive complete response or partial response after induction therapy will receive lenalidomide 25 mg qd po during 1-10 days in every 21 days for 2 years.
  Arms: ZR2

SUMMARY:
A multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of Pola-ZR2 (polatuzumab vedotin, zanubrutinib, rituximab and lenalidomide) versus ZR2 (zanubrutinib, rituximab and lenalidomide) in the treatment of old patients with de novo diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of Pola-ZR2 versus ZR2 in the treatment of elderly de novo diffuse large B-cell lymphoma patients. Subjects will be randomly assigned 1:1 to Pola-ZR2 or ZR2 regimen. The stratification will be performed according to international prognostic index (2-3 / 4-5).

Patients in Pola-ZR2 group will receive 6 cycles of polatuzumab vedotin 1.8 mg/kg, day 2 on the 1st cycle and day 1 on the 2nd to 6th cycle, zanubrutinib 160mg bid, day 1-21, orally, lenalidomide 25mg qd, day 2-11, orally, rituximab 375mg/m², day 1, intravenously, every 21 days. Patients in ZR2 group will receive 6 cycles of zanubrutinib 160mg bid, day 1-21, orally, lenalidomide 25mg qd, day 2-11, orally, rituximab 375mg/m², day 1, intravenously, every 21 days.

Patients who receive complete response or partial response after induction therapy will receive lenalidomide 25 mg qd po during 1-10 days in every 21 days for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following criteria to be enrolled in the study:

* Histologically-confirmed diffuse large B-cell lymphoma (without central nervous system involvement)
* Aged ≥ 80 years old or aged 70-79 with comprehensive geriatric assessment stratified as unfit or frail
* International prognostic index score 2 to 5
* At least 1 measurable site of disease (defined as lymph nodes with the long diameters longer than 1.5cm, or extra-nodal sites with the long diameters longer than 1.0cm; meanwhile, any lesion site with at least 2 measurable vertical diameters)
* Able to swallow capsules
* Life expectancy of at least 3 months determined by researchers
* The patient or his or her legal representative must provide written informed consent prior to any special examination or procedure for the research.
* Anti-lymphoma drugs have not been used before (except glucocorticoids)

Exclusion Criteria:

Presence of any of the following criteria will exclude a patient from enrollment:

* Uncontrolled blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

Neutrophils<1.5×10^9/L Platelets<80×10^9/L ALT or AST is 2 times higher than the upper limits of normal (ULN), serum bilirubin are 1.5 times higher than the ULN.

Creatinine is 1.5 times higher than the ULN or eGFR is lower than 40ml/min/1.73m^2 (according to Cockcroft-Gault Equation or MDRD Equation).

* uncontrollable or significant cardiovascular diseases, including but not limited to: Left ventricular ejection fraction<50% Cardiomyopathy, such as dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy QTc prolongation with clinical significance, QTc interval>470ms (females) or 480ms (males), type 2 second-degree atrioventricular block or third-degree atrioventricular block
* Patients with HbsAg positive are required to have HBV DNA<1.0×10^3 IU/ml before entering the group. In addition, if the patient is HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA test is also required, and HBV DNA<1.0×10^3 IU/ml is required before entering the group
* Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
* HIV-infected patients
* History of stroke or intracranial hemorrhage within 6 months prior to start of therapy
* Other medical conditions determined by the researchers that may affect the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2028-08-10 (Estimated); Study Completion 2029-08-10 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | up to approximately 2 years

SECONDARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
2-year OS rate | Baseline up to data cut-off (up to approximately 2 years)
  2-year OS rate
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Complete response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Overall response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]]
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 5 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Percentage of Participants Achieving Meaningful Improvement in European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by EORTC QLQ-C30 (Verison 3.0).
Percentage of Participants Achieving Meaningful Improvement in EORTC QLQ-ELD14 (Elderly Module) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by EORTC QLQ-ELD14.
Percentage of Participants Achieving Meaningful Improvement in Functional Assessment of Cancer Therapy-Lymphoma Lymphoma Subscale (FACT-Lym LymS) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by FACT-Lym LymS.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Hematology, Rui-Jin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No